CLINICAL TRIAL: NCT06568341
Title: Turkish Validity and Reliability of the Outcome Expectations For Yoga Scale
Brief Title: Turkish Validity-Reliability of the Outcome Expectations For Yoga Scale
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Muzeyyen Oz, Research Assistant, PhD, Principal Investigator, Hacettepe University
Other Study IDs: 8931c5a6b0c54418
Record Dates: First submitted 2024-08-16; First posted 2024-08-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Adults
Keywords: yoga; outcome expectations; psychometric; validation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: validity and reability study — Validity and reliability assessment of the Turkish version of the Outcome Expectations For Yoga (OEY) Scale

SUMMARY:
Evaluation of the Turkish validity and reliability of the outcome Expectations for Yoga (OEY) Scale, which was developed to evaluate attitudes and beliefs related to yoga practice

DETAILED DESCRIPTION:
The Turkish version of the Outcome Expectations for Yoga (OEY) scale will be studied. The OEY scale is designed to assess the physical, mental, and spiritual health benefits associated with yoga practice in adults.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older

Exclusion Criteria:

* Pregnant women
* Body Mass Index above 40
* Practiced yoga, Tai Chi, Qi Gong, or a mindfulness-based therapy program 2 times or more in the past month or 10 times in the past year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 years and older
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The Outcome Expectations for Yoga (OEY) Scale | 6 months
  Reliability and Validity of OEY scale by Correlation Analysis.

SECONDARY OUTCOMES:
Five Facet Mindfulness Questionnaire Short Form | 6 months
  Individuals' mindfulness levels will be evaluated. The scale evaluates individuals' mindfulness levels under 5 factors ("Observing", "Describing", "Acting with Awareness", "Non-Judgement", and "Non-Reactivity"). A 5-point Likert-type assessment (1=Never, 2=Rarely, 3=Sometimes, 4=Frequently, 5=Almost Always) is used in the evaluation of scale items. Higher scores are indicative of someone who is more mindful in their everyday life.
Exercise Self Efficacy Scale | 6 months
  Individuals' exercise self-efficacy will be assessed. The Exercise Self-Efficacy Scale consists of 6 questions scored between 0-100 (0=not confident at all, 100=completely confident) on a visual analog scale and measures the self-efficacy of individuals to exercise despite various barriers. The total score is obtained by summing the scores of the 6 questions. As the score increases, the level of self-efficacy also increases.
International Physical Activity Questionnaire-Short Form | 6 months
  Physical activity levels of individuals will be evaluated.
Short Form-12 Health Survey | 6 months
  Individuals' quality of life will be assessed. Short Form-36 is a 36-item self-reported test developed to measure eight different health concepts (physical functioning, social functioning, role limitations due to physical problems, role limitations due to emotional problems, mental health, energy/fatigue, bodily pain, and general health perception) in any general or clinical population. Short Form-12 is a shorter version of Short Form-36 and includes the same sub-dimensions. The scale can be scored between 0-100. Higher scores indicate higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem Ulger, Prof, Study Director — Hacettepe University
Locations (2):
- Turkey (Türkiye) (2):
  - Hacettepe University Faculty of Physical Therapy and Rehabilitation, Ankara, Altindag
  - Çankiri Karatekin University, Çankırı

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thind H, Sillice MA, Fava JL, Lantini R, Horowitz S, Jennings E, Rosen RK, Carmody J, Becker BM, Marcus BH, Bock BC. Development and Validation of the Outcome Expectations for Yoga Scale. Am J Health Behav. 2017 Nov 1;41(6):796-802. doi: 10.5993/AJHB.41.6.13. PMID 29025507
- [Background] Resnick B, Zimmerman SI, Orwig D, Furstenberg AL, Magaziner J. Outcome expectations for exercise scale: utility and psychometrics. J Gerontol B Psychol Sci Soc Sci. 2000 Nov;55(6):S352-6. doi: 10.1093/geronb/55.6.s352. PMID 11078112
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735